CLINICAL TRIAL: NCT05677464
Title: Prospective Multicenter Study to Assess the Safety and Efficacy of the Endomina® Triangulation Platform for Treating Patients Requiring Endoscopic Gastroplasty
Brief Title: Prospective Multicenter Study With the Endomina® Triangulation Platform
Acronym: PRETTi
Status: Recruiting | Type: Observational
Sponsor: Endo Tools Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: ST-2019-001
Record Dates: First submitted 2022-12-23; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Obesity
Keywords: Obesity; Gastroplasty; Endoscopic gastroplasty; endomina
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This registry is designed to further assess on a larger scale safety and efficacy of the endomina® device and tissue apposition accessories (TAPES) when used in the frame of "real life" routine clinical practice

DETAILED DESCRIPTION:
This is a single arm prospective, multi-center international, open-label, non-interventional, , post-market study. This registry is designed to further assess on a larger scale safety and efficacy of the endomina® and TAPES devices. Patients in need of endoscopic gastroplasty will be enrolled and followed-up for 36 months following hospital routine practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be willing to provide written informed consent
* Adult patients (between ≥ 18 years (legal age in Europe) and 65 years of age at time of ESG)
* Patients who require endoscopic gastroplasty and who are selected by multidisciplinary team/investigators to be treated with the endomina® device and accessories according to the Instructions for Use (IFU)

Exclusion Criteria:

* Patients with impaired hemostasis or pre-existing conditions that may lead to fragile mucosa (i.e., any contraindication to suturing the stomach)
* Any malformation from mouth to esophagus (including pharynx)
* Any contraindication to general anesthesia, including patients with cardiorespiratory dysfunction or respiratory failure
* Woman who are pregnant, at the time of the procedure or planning (trying) to become pregnant, or nursing within 12 months after the procedure.
* Impending surgery 60 days post intervention of the treated section of the GI tract
* Participation in another clinical study evaluating another medical device, another procedure or a medication that did not reach its primary endpoint

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients, who require endoscopic gastroplasty (ESG) and who are selected by multidisciplinary team/investigators to be treated with the endomina® device.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety outcome | 12 months
  Occurrence of Serious Adverse Device Effects at 12 months.
Technical success | 1 day
  Technical success defined by the completion of the intended procedure without premature abortion due to technical reasons/device deficiency

CONTACTS AND LOCATIONS:
Overall Officials: Mrs Leclercq, Study Director — Endo Tools Therapeutics S.A.
Locations (1):
- Endo Tools Therapeutics S.A., Gosselies, Wallonia, Belgium

IPD SHARING:
Plan to Share IPD: Undecided